CLINICAL TRIAL: NCT05596045
Title: A Phase Ib, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability, Efficacy and Pharmacokinetics of ASC10 Tablets in Mild or Moderate COVID-19 Patients
Brief Title: Study to Evaluate Safety, Tolerability, Efficacy and Pharmacokinetics of ASC10 in Mild to Moderate COVID-19 Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study has been cancelled due to business reasons.
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC10-102
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2022-10

CONDITIONS: SARS CoV 2 Infection
Keywords: ASC10; RdRp
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASC10 (Experimental): Participants will be randomized to receive 200, 400 and 800 mg ASC10 BID for 5.5 days
  Interventions: Drug: ASC10
- Placebo (Placebo Comparator): Participants will be randomized to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC10 — Participants will be randomized to receive 200, 400 and 800 mg ASC10 BID for 5.5 days
  Arms: ASC10
Drug: Placebo — Participants will be randomized to receive placebo
  Arms: Placebo

SUMMARY:
This is a phase Ib, randomized, double-blind, placebo-controlled study to evaluate safety, tolerability, efficacy and pharmacokinetics of ASC10 tablets in mild or moderate COVID-19 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years at screening;
2. Those females who do not have plans for pregnancy within six months and are willing to take effective contraceptive measures from the first dose of the study drug to 3 months after the last dose;
3. If male, agree to use adequate contraception throughout the study and for at least 3 months after the last dose of study drug;
4. Has a documentation of PCR-confirmed SARS-CoV-2 infection with sample collection ≤5 days prior to randomization.

Exclusion Criteria:

1. Females who are pregnant, planning to become pregnant, or breastfeeding;
2. Has at least one characteristic or underlying medical condition associated with an increased risk of developing severe or critical illness from COVID-19;
3. Has hypersensitivity or other contraindication to any of the components of the study interventions;
4. Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-28 (Estimated); Primary Completion 2023-03-08 (Estimated); Study Completion 2023-10-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Event (TEAEs) in multiple ascending doses | From Day 0 to Study Completion, up to 32 days
PK parameters for ASC10, GLC01-700 (molnupiravir) and ASC10-A in plasma as AUC0-12h | From Day 1 to Day 6

SECONDARY OUTCOMES:
Time (days) to sustained resolution of all targeted COVID-19 signs/symptoms | From Day 1 to Study Completion, up to 32 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pinnacle Research Group, Anniston, Alabama
  - Aga Clinical Trials, Hialeah, Florida